CLINICAL TRIAL: NCT00886886
Title: Pharmacological Interaction Between Reboxetine and 3,4-Methylenedioxymethamphetamine (MDMA, Ecstasy): Pharmacological Effects and Pharmacokinetics
Brief Title: Interaction Between Reboxetine and 3,4-Methylenedioxymethamphetamine: Pharmacodynamics (PD) and Pharmacokinetics (PK)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: EKBB373/08
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Mood Disorder; Substance-related Disorders; Amphetamine-related Disorders
Keywords: MDMA; norepinephrine; Ecstasy; stimulant
MeSH Terms: conditions — Mood Disorders; Substance-Related Disorders; Amphetamine-Related Disorders | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Reboxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Reboxetine, MDMA, Placebo (Other): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 1 arm but two (actually 4) treatment conditions in the same subject.
  Interventions: Drug: MDMA; Drug: Reboxetine, 8 mg; Drug: Placebo

INTERVENTIONS:
Drug: MDMA — 125 mg, single dose
Drug: Reboxetine, 8 mg — two doses 12h and 2h before MDMA
Drug: Placebo — capsules identical to MDMA or Reboxetine

SUMMARY:
MDMA releases dopamine, serotonin, and norepinephrine in the brain. Serotonin uptake inhibitors have been shown to interact with 3,4-Methylenedioxymethamphetamine (MDMA) and to decrease its psychoactive and cardiovascular stimulant effects. This finding indicates that MDMA acts in part by releasing serotonin through the serotonin uptake site. However, in vitro studies show that MDMA binds more potently to the norepinephrine uptake site that to the the serotonin or dopamine uptake transporter. In addition, norepinephrine uptake site blockers such antidepressant drugs attenuate some of the behavioral effects of MDMA in animals. These preclinical data indicate that norepinephrine may also contribute to the response to MDMA in humans. To test this hypothesis this study evaluates the interacting effects of the selective norepinephrine transporter inhibitor reboxetine on the subjective and cardiovascular stimulant effects of MDMA in healthy volunteers.

DETAILED DESCRIPTION:
The study will use a randomized double-blind cross-over design with four experimental sessions. Reboxetine (8 mg) or placebo will be administered the night before the experimental session and 1 h before the administration of MDMA (125 mg) or placebo to 16 healthy volunteers. Subjective and cardiovascular responses and plasma samples for pharmacokinetics will be repeatedly assessed throughout the experiments.

We hypothesize that the highly selective norepinephrine uptake inhibitor reboxetine will attenuate subjective and especially heart rate and blood pressure responses to MDMA. Such a result would indicate that norepinephrine is critically involved in the pharmacology of MDMA and may provide helpful in the use and development of treatments for Ecstasy intoxications.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient understanding of the German language
* Subjects understand the procedures and the risks associated with the study
* Participants must be willing to adhere to the protocol and sign the consent form
* Participants must be willing to refrain from taking illicit psychoactive substances during the study.
* Participants must be willing to drink only alcohol-free liquids and no xanthine-containing liquids (such as coffee, black or green tea, red bull, chocolate) after midnight of the evening before the study session. Subjects must agree not to smoke tobacco for 1 h before and 4 hours after MDMA administration.
* Participants must be willing not to drive a traffic vehicle in the evening of the study day.
* Women of childbearing potential must have a negative pregnancy test at the beginning of the study and must agree to use an effective form of birth control. Pregnancy tests are repeated before each study session.
* Body mass index: 18-25 kg/m2

Exclusion Criteria:

* Chronic or acute medical condition including clinically relevant abnormality in physical exam, laboratory values, or ECG. In particular: Hypertension (>140/90 mmHg). Personal or first-grade history of seizures. Cardiac or neurological disorder.
* Current or previous psychotic or affective disorder
* Psychotic or affective disorder in first-degree relatives
* Prior illicit drug use (except Tetrahydrocannabinol-containing products) more than 5 times or any time within the previous 2 months.
* Pregnant or nursing women.
* Participation in another clinical trial (currently or within the last 30 days)
* Use of medications that are contraindicated or otherwise interfere with the effects of the study medications (monoamine oxidase inhibitors, antidepressants, sedatives etc.)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Effect of reboxetine on subjective responses to MDMA | 24h

SECONDARY OUTCOMES:
Effect of reboxetine on physiological responses to MDMA | 24h
Effects of reboxetine on pharmacokinetics of MDMA | 24h
Tolerability of MDMA and reboxetine | 7 days
Effect of reboxetine on neuroendocrine responses to MDMA | 24h

OTHER OUTCOMES:
Genetic polymorphisms | assessed after study completion
  Effects of genetic polymorphisms on the response to MDMA

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, Principal Investigator — Department of Internal Medicine, Division of Pharmacology & Toxicology, University Hospital Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland

REFERENCES:
- [Derived] Vizeli P, Liechti ME. Oxytocin receptor gene variations and socio-emotional effects of MDMA: A pooled analysis of controlled studies in healthy subjects. PLoS One. 2018 Jun 18;13(6):e0199384. doi: 10.1371/journal.pone.0199384. eCollection 2018. PMID 29912955
- [Derived] Hysek CM, Liechti ME. Effects of MDMA alone and after pretreatment with reboxetine, duloxetine, clonidine, carvedilol, and doxazosin on pupillary light reflex. Psychopharmacology (Berl). 2012 Dec;224(3):363-76. doi: 10.1007/s00213-012-2761-6. Epub 2012 Jun 15. PMID 22700038